CLINICAL TRIAL: NCT02033863
Title: PrOspective, MultiCenter Study for the Evaluation of PerformanCe of the ArtVentive Medical Group Peripheral EndoLuminal OcclUsion SystemTM in the Treatment of Varicocele or Pelvic Congestion SynDromE - OCCLUDE I
Brief Title: Evaluation of PerformanCe of the Peripheral EOS in the Treatment of Varicocele or Pelvic Congestion SynDromE
Acronym: OCCLUDE-I
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ArtVentive Medical Group, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TD 0080/07
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Varicocele; Pelvic Congestion Syndrome
Keywords: Varicocele; Pelvic Congestion Syndrome; Pelvic Venous Incompetence; Ovarian Varices
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: Varicocele arising from the spermatic vein(s) and pampiniform plexus, with or without concomitant diagnosis of infertility or subfertility
- Cohort B: Pelvic varices in females for the treatment of pelvic congestion syndrome (e.g., pelvic venous incompetence).

SUMMARY:
To collect confirmatory data in support of the safety and performance of the ArtVentive Medical Group Endoluminal Occlusion System.

DETAILED DESCRIPTION:
Prospective, non-randomized, multi-center confirmatory observational study for the treatment of subjects with the need for vascular occlusion for the following conditions:

1. Cohort A: Varicocele arising from the spermatic vein(s) and pampiniform plexus, with or without concomitant diagnosis of infertility or subfertility
2. Cohort B: Pelvic varices in females for the treatment of pelvic congestion syndrome (e.g., pelvic venous incompetence).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥18 to ≤75 years.
2. Subject with target vessels of 3.0 mm to 12.0 mm in diameter.
3. Subject having indications to undergo embolotherapy consistent with clinical and pre-procedural angiographic assessment for spermatic vein origin varicocele (unilateral and/or bilateral) or pelvic congestion syndrome (pelvic venous incompetence).
4. Subject is able and willing to comply with site standard medical follow-up, including one month follow-up visit.
5. Subject or subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the consent form.

Exclusion Criteria:

1. Subject has an active systemic infection.
2. Subject has a known allergy to iodinated contrast for which they cannot be adequately premedicated.
3. Subject has history of stroke within the prior 6 months.
4. Subject has history of myocardial infarction with the prior 3 months.
5. Subject has acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L), or on dialysis.
6. Subject has a known coagulopathy or has a bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter, or INR >1.5.
7. Co-morbid conditions that place the subject at an unacceptable surgical risk (e.g., severe chronic obstructive pulmonary disease, hepatic failure, cardiac disease, autoimmune disorders or conditions of severe immunosuppression).
8. Subjects in whom venography or arteriography is contraindicated.
9. Subjects with known hypersensitivity or contraindication to nickel or nitinol.
10. Subject has a less than one year life expectancy.
11. Subject is pregnant or breastfeeding.
12. Subject with endometriosis or other ovarian / uterine pathology with adhesions that would interfere with the endpoints of this study.
13. Subject with previous pelvic surgical intervention or embolotherapy for varicocele or ovarian varices that would interfere with the endpoints of this study, including but not limited to, recurrent varicocele or ovarian varices.
14. Any clinical evidence that the investigator feels would place the subject at increased risk with the deployment of the device.
15. Subject has planned concomitant procedure at the time of the embolization (e.g., coil embolization, etc.).
16. Subject is participating in another study of a device, medication, biologic, or other agent within 30 days or could, in the opinion of the investigator, impact the results of this study.
17. Subject has other medical, social or psychological problems that in the opinion of the investigator would preclude them from receiving this treatment and the procedures and or participating in evaluations pre- and post-treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring permanent occlusion of the peripheral vessels for the following conditions:
  1. Cohort A: Varicocele arising from the spermatic vein(s) and pampiniform plexus, with or without concomitant diagnosis of infertility or subfertility.
  2. Cohort B: Pelvic varices in females for the treatment of pelvic congestion syndrome (e.g., pelvic venous incompetence).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Safety | Acute & 30 days
  Composite of new-onset major device-related adverse event(s) including device embolization beyond targeted treatment area (not therapeutic indication of embolization), need for emergency surgical intervention of the target vessel, or distal embolization (non-device embolization, e.g., particulate matter / plaque distal to the device) at 30 days.

SECONDARY OUTCOMES:
Pain | Acute & 30 days
  Reduction of pain.
Recurrent varices | 30 days
  Recurrence of varices requiring repeat embolizations within 30 days.
Occlusion | 30 days
  Sustained occlusion at 30 days follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Maleux, MD, Principal Investigator — UZ Leuven, Belgium
Locations (3):
- UZ Leuven, Leuven, Belgium
- University Hospital No4, Lubin, Poland
- Ospedale Regionale di Lugano, Lugano, Switzerland

REFERENCES:
- [Background] Venbrux AC, Rudakov L, Plass A, Emmert MY, Ebner A. A new occlusion device: application of the ArtVentive endoluminal occlusion system (EOS)--first in human clinical trial. Cardiovasc Intervent Radiol. 2014 Feb;37(1):85-93. doi: 10.1007/s00270-013-0626-y. Epub 2013 May 24. PMID 23703667